CLINICAL TRIAL: NCT00053521
Title: Genetic Epidemiology of CVD Risk Factors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1206; R01HL070167-01 (NIH); R01HL069995-01 (NIH)
Record Dates: First submitted 2003-01-30; First posted 2003-01-31 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine the role of genetic factors influencing risk factors for cardiovascular disease, ultimately identifying specific genes influencing the age-related progression of cardiovascular disease risks.

DETAILED DESCRIPTION:
BACKGROUND:

Understanding the genetic basis of common multifactorial diseases such as cardiovascular disease (CVD) remains an elusive goal, but the great advances in molecular genetic technology, statistical genetic methods, and phenotypic assessment of CVD risk factors in recent years have facilitated more sophisticated genetic studies of risks for heart disease.

The study is a follow-up to one conducted in the 1970's and 1980's. The availability of 5 large kindreds first identified and recruited as part of the "High Blood Pressure in the Young" program is an important resource. The investigators have an extensive array of baseline data that was collected in the late 1970s and early 1980s on 750 participants stemming from that project, although some data are available only on a subset of participants. The present study population centers on 764 individuals in five large, multigenerational, extended families (four white and one African-American) originally examined 25 years ago. Data collected from the original participants include hundreds of biochemical, medical, physiological, behavioral, physical, psychological, genetic and demographic traits.

DESIGN NARRATIVE:

The study consists of four specific aims: 1) Collect 25-year follow-up data from approximately 500 of the original participants, and new data from approximately 500 of their relatives not examined in the original study. The cardiovascular disease risk factor phenotypes to be collected include hemodynamic measures, carotid intima-media thickness, and measures of cardiopulmonary function. 2) Obtain DNA samples from these 1,000 individuals and use modern high-throughput molecular genotyping methods to create a 10 cM genetic marker map. 3) Quantify and characterize the nature of genetic influences on CVD risk factors using quantitative genetic methods suited for cross-sectional and serial (follow-up) data from relatives in large extended families. 4) Conduct linkage analyses to identify chromosomal regions (QTLs) harboring genes that influence individual variation in cardiovascular disease risk factors. Following these linkage analyses, the investigators will examine more closely the strongest linkage signals with fine mapping linkage analysis in order to narrow chromosomal regions of interest. The study is a collaboration between Wright State University and the Southwest Foundation for Biomedical Research.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Cole — Southwest Foundation for Biomedical Research; Roger Siervogel — Wright State University